CLINICAL TRIAL: NCT03199001
Title: Native T1 Mapping by Cardiovascular Magnetic Resonance Imaging in Rare Diseases- A New Method to Improve Patient Care
Brief Title: Native T1 Mapping by Cardiovascular Magnetic Resonance Imaging in Rare Diseases
Acronym: FABRY400
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Collaborators: University Hospital Birmingham (Other); University of Sydney (Other)
Responsible Party: Sponsor
Other Study IDs: 14/0354
Record Dates: First submitted 2017-06-19; First posted 2017-06-26 (Actual); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Fabry Disease
Keywords: Fabry Disease; T1 Mapping; Cardiovascular Magnetic Resonance
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma and urine samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Fabry Disease (FD) is a rare, X-linked lysosomal storage disorder leading to left ventricular hypertrophy, myocardial fibrosis, arrhythmia and heart failure. Cardiac involvement is the leading cause of death in FD. Treatment with enzyme replacement therapy is expensive, may be poorly targeted and there are difficulties in early detection and disease monitoring. T1 mapping signal change is a potential remarkable biomarker for FD.

Fabry400 is a multicentre study aiming to understand the biology of Fabry Disease and its relationship to non-invasive multi parametric mapping by CMR.

DETAILED DESCRIPTION:
Our understanding of cardiac involvement in FD is limited because the myocyte storage cannot be assessed non-invasively. However with the development of CMR T1 mapping this maybe possible. T1 mapping demonstrated excellent discrimination between FD and other causes of LVH, and this property is highly suggestive of a direct but intricate relationship between T1 signals and abnormal fat storage. Specifically, 50% of patients without LVH have low T1 values, suggesting that T1 is an early disease marker in FD. This property may prove particularly useful for assessing disease progression and treatment response in early disease.

In CMR, LGE in FD characteristically occurs in the basal inferolateral wall. LGE is associated with a poor response to therapy and adverse outcomes. Hybrid imaging with PET/MR has shown that some FD LGE may be inflammation. T2 mapping may be useful as it is a sensitive detector of inflammation and oedema, for example discriminating acute from chronic myocardial infarction, and diagnosing myocarditis, particularly in the setting of chronic myocarditis or heart failure.

The aims of this study are:

1. Improve the diagnosis of cardiac involvement by recognition of early disease
2. Detect early changes and responses to therapy
3. Improve the understanding of the pathophysiology of cardiac involvement using multiparametric mapping by CMR

Study Method:

This is a cohort observational study of FD patients including children, patients starting ERT, ERT naïve patients and LVH positive patients. Follow up scans at 6 months and 12 months will be done on patients starting ERT. CMR Scanning will use T1 and T2 mapping techniques against established gold-standard sequences. The patients will also have ECHO and ECG. Blood biomarkers will be collected (serum, plasma and urine).

ELIGIBILITY:
Inclusion Criteria:

* Gene-positive Fabry Disease
* Male or female
* Age at least 9 years

Exclusion Criteria:

* Any absolute contraindication to CMR
* Pregnancy

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Fabry Disease patients recruited from Fabry outpatient clinics
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2015-02-19 (Actual); Primary Completion 2018-08-19 (Estimated); Study Completion 2019-02-19 (Estimated)

PRIMARY OUTCOMES:
Presence of storage in Fabry cardiomyopathy | 1 hour
  Presence or absence of storage (measured in milliseconds) by T1 mapping by CMR

SECONDARY OUTCOMES:
Presence of inflammation in Fabry cardiomyopathy | 1 hour
  Presence or absence of inflammation (measured in milliseconds) by T2 mapping by CMR
Change in storage measure | 12 months
  Change in storage measure (measured in milliseconds) by T1 mapping by CMR

CONTACTS AND LOCATIONS:
Locations (4):
- University of Sydney, Sydney, Australia
- United Kingdom (3):
  - University Hospital Birmingham, Birmingham
  - Royal Free Hospital, London
  - The Heart Hospital, University College London Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sado DM, White SK, Piechnik SK, Banypersad SM, Treibel T, Captur G, Fontana M, Maestrini V, Flett AS, Robson MD, Lachmann RH, Murphy E, Mehta A, Hughes D, Neubauer S, Elliott PM, Moon JC. Identification and assessment of Anderson-Fabry disease by cardiovascular magnetic resonance noncontrast myocardial T1 mapping. Circ Cardiovasc Imaging. 2013 May 1;6(3):392-8. doi: 10.1161/CIRCIMAGING.112.000070. Epub 2013 Apr 5. PMID 23564562
- [Background] Pica S, Sado DM, Maestrini V, Fontana M, White SK, Treibel T, Captur G, Anderson S, Piechnik SK, Robson MD, Lachmann RH, Murphy E, Mehta A, Hughes D, Kellman P, Elliott PM, Herrey AS, Moon JC. Reproducibility of native myocardial T1 mapping in the assessment of Fabry disease and its role in early detection of cardiac involvement by cardiovascular magnetic resonance. J Cardiovasc Magn Reson. 2014 Dec 5;16(1):99. doi: 10.1186/s12968-014-0099-4. PMID 25475749
- [Background] Nappi C, Altiero M, Imbriaco M, Nicolai E, Giudice CA, Aiello M, Diomiaiuti CT, Pisani A, Spinelli L, Cuocolo A. First experience of simultaneous PET/MRI for the early detection of cardiac involvement in patients with Anderson-Fabry disease. Eur J Nucl Med Mol Imaging. 2015 Jun;42(7):1025-31. doi: 10.1007/s00259-015-3036-3. Epub 2015 Mar 26. PMID 25808629
- [Derived] Cheepvasarach C, Gribble M, Ugander M, Vijapurapu R, Nordin S, Augusto J, Steeds RP, Tchan M, Moon JC, Pathan F, Kozor R. Left atrial strain tracks abnormal ventricular mechanics in Fabry disease. Open Heart. 2025 Oct 31;12(2):e003385. doi: 10.1136/openhrt-2025-003385. PMID 41176334
- [Derived] Vijapurapu R, Nordin S, Baig S, Liu B, Rosmini S, Augusto J, Tchan M, Hughes DA, Geberhiwot T, Moon JC, Steeds RP, Kozor R. Global longitudinal strain, myocardial storage and hypertrophy in Fabry disease. Heart. 2019 Mar;105(6):470-476. doi: 10.1136/heartjnl-2018-313699. Epub 2018 Oct 3. PMID 30282640